CLINICAL TRIAL: NCT04352257
Title: Bladder and Prostate Sonomorphology as a Useful Tool for Detecting Bladder Outlet Obstruction in Patients With Symptomatic Benign Prostatic Hyperplasia
Brief Title: Bladder and Prostate Sonomorphology in Patients With Symptomatic Benign Prostatic Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Diaa Eldin Taha Ramadan Mohamed, Lecturer of urology, Kafrelsheikh University
Other Study IDs: RS/19.21
Record Dates: First submitted 2020-04-12; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasonography: pelvic and transrectal ultrasound
  Interventions: Radiation: pelvic Ultrasound

INTERVENTIONS:
Radiation: pelvic Ultrasound — pelvic and transrectal ultrasound
  Other Names: transrectal ultrasound

SUMMARY:
Bladder and Prostate Sonomorphology in Patients With Symptomatic Benign Prostatic Hyperplasia?

DETAILED DESCRIPTION:
Bladder and Prostate Sonomorphology as a Useful tool for Detecting Bladder Outlet Obstruction in Patients With Symptomatic Benign Prostatic Hyperplasia?

ELIGIBILITY:
Inclusion Criteria:

male patients with LUTS/BPH prostate size > 25 g

Exclusion Criteria:

urinary retention diabetes mellitus neurologic deficit LUTS medications prior lower urinary tract surgery concomitant bladder pathology small bladder capacity (< 150 ml) urethral stricture evident prostate carcinoma.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient more than 50 year old who were presented with Lower urinary tract symptoms.The patients were be subjected to pelvic and transrectal ultrasound.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
pelvic and transrectal ultrasound | 18 months
  bladder wall thickness, prostate volume, and prostate morphology

SECONDARY OUTCOMES:
pelvic and transrectal ultrasound in relation to pressure flow study | 18 months
  correlation of the pelvic and transrectal ultrasound parameters to pressure flow study measurements

CONTACTS AND LOCATIONS:
Overall Officials: Diaa Eldin Taha, MD, Principal Investigator — Lecturer of urology
Locations (1):
- Kafrelsheikh faculty of medicine, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No